CLINICAL TRIAL: NCT00736307
Title: Transplantation of Ex-Vivo Expanded Human Limbal Epithelial Stem Cells (LSC) on Amniotic Membrane (AM) for Limbal Stem Cell Deficiency (LSCD)
Brief Title: Autologous Transplantation of Cultivated Limbal Stem Cells on Amniotic Membrane in Limbal Stem Cell Deficiency (LSD) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Collaborators: Small Business Developing Center (Unknown); Labafi Nejad Eye Research Center (Unknown)
Responsible Party: Hamid Gourabi/ Chief, Royan Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROYAN-EYE-001
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2010-04

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: limbal stem cell deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cultured limbal stem cells Transplantation
  Interventions: Procedure: Cultured limbal stem cells Transplantation

INTERVENTIONS:
Procedure: Cultured limbal stem cells Transplantation — Transplantation of cultivated limbal epithelium on amniotic membrane
  Other Names: Transplantation

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and long term outcomes of ex vivo cultured limbal stem cell on amniotic membrane transplantation for corneal surface reconstruction in cases of partial and sever limbal stem cell deficiency.

DETAILED DESCRIPTION:
Ocular surface is composed of corneal and conjunctival epithelial cells. Normal cornea is essential for normal vision. Defects in renewal and repair of ocular surface as a result of limbal stem cell deficiency are now known to cause varying ocular surface morbidity including persistent photophobia, repeated and persistent surface breakdown and overt conjunctivalisation of the cornea. Restoring ocular health in these eyes has traditionally been frustrating. Ex vivo cultured limbal epithelial stem cells have been used successfully to treat limbal stem cell deficiency. Ex-vivo limbal stem cell allograft transplantation is achieved by harvesting limbal corneal tissue from donor eyes (either matched living relatives or cadaveric donors). The donor stem cells are obtained by excising a small area of the conjunctiva at the limbus and are a minor procedure. The tissue so obtained is then grown in tissue culture and once the cells have multiplied sufficiently, small sheets are transplanted on to the affected eye(s), backed with an amniotic membrane. The surgery is undertaken under either local or general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unilateral limbal stem cell insufficiency and totally corneal vascularization
* Presence of Goblet cells on the cornea
* Minimum tear was about 5 mm
* Minimum duration of deficiency was 3 years
* Vision was Light Perception

Exclusion Criteria:

* Systemic disease affecting both eyes such as Stevens-Johnson syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Snellen visual acuity | 6 months
corneal epithelial integrity and stability | 6 months

SECONDARY OUTCOMES:
Impression cytology | 12 months
Extent of retarding recurrent neovascularisation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gorabi, PhD, Study Chair — Royan institute, Tehran, Iran; Mohammadali Javadi, MD, Study Chair — Labbafinejad Ophthalmic Research Center, Tehran, Iran; Hossein Baharvand, PhD, Principal Investigator — Royan institute, Tehran, Iran; Alireza Baradaran, MD, Principal Investigator — Labbafinejad, Ophthalmic Research Center, Tehran, Iran; Marzieh Ebrahimi, PhD, Study Director — Royan Institute, Tehran, Iran
Locations (2):
- Iran (2):
  - Royan Institute, Tehran, Tehran Province
  - Labbafinejad Ophthalmic Research Center, Tehran, Tehran Province

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org